CLINICAL TRIAL: NCT01164189
Title: Randomized Trial Assessing the Significance of Bevacizumab in Recurrent Grade II and Grade III Gliomas - The TAVAREC Trial
Brief Title: Bevacizumab in Recurrent Grade II and III Glioma
Acronym: TAVAREC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26091; 2009-017422-39 (EudraCT Number)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult pineal gland astrocytoma; adult subependymal giant cell astrocytoma; adult oligodendroglioma; adult anaplastic oligodendroglioma; recurrent adult brain tumor; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Brain Neoplasms; Glioblastoma; Gliosarcoma; Glioma | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temozolomide (Other): Administered orally on day 1-5, 150-200 mg/m(2), repeated every 4 weeks, up to 12 cycles
  Interventions: Drug: Temozolomide
- Temozolomide + Bevacizumab (Experimental): TMZ: Administered orally on day 1-5, 150-200 mg/m(2), repeated every 4 weeks, up to 12 cycles
  Beva: 10 mg/kg bw IV in 90 minutes on day 1 and 14, 4 week cycles.
  Interventions: Biological: Bevacizumab; Drug: Temozolomide

INTERVENTIONS:
Biological: Bevacizumab — Bevacizumab (vial of 400mg/16mL) at a dose of 10 mg/kg bodyweight i.v. in 90 min on day 1 and day 14 of 4 week cycles
  Other Names: Avastin
  Arms: Temozolomide + Bevacizumab
Drug: Temozolomide — Temozolomide (250, 100, 20 and 5 mg caps) will be administered orally on day 1-5, 150-200 mg/m², and will be repeated every 4 weeks. This will be repeated for up to 12 cycles.
  Other Names: Temodar; Temodal; Temcad

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether temozolomide is more effective when given with or without bevacizumab in treating patients with recurrent glioma.

PURPOSE: This randomized clinical trial is studying how well temozolomide works with or without bevacizumab in treating patients with recurrent glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To document the activity of both combination temozolomide plus bevacizumab and temozolomide alone in patients with recurrent grade II or grade III glioma without 1p/19q co-deletion.

Secondary

* To characterize the safety of treatment in these patients.
* To document the quality of life and cognitive functioning, as a measure of clinical benefit, of these patients.
* To explore qualification or occurrence of prognostic and/or predictive biomarkers of activity or efficacy in these patients. (exploratory)
* To document the discordances between RANO and Macdonald's criteria for the evaluation of response and progression. (exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to institution, initial histology (grade II vs grade III), WHO performance status (0-1 vs 2), and prior treatment (radiotherapy [RT] alone, temozolomide [TMZ] or procarbazine, lomustine and vincristine [PCV] alone vs TMZ/RT). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral temozolomide as in arm I and bevacizumab IV over 90 minutes on days 1 and 15. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

Patients complete neurocognitive questionnaires (i.e., the Hopkins Verbal Learning test, the Controlled Oral Word Association test, and the Trail Making tests A and B). Quality-of-life assessment questionnaires, including EORTC QLQ-C30 and EORTC-BN20, are completed by both patients and caregivers/relatives at baseline and then periodically.

Frozen tumor biopsies or paraffin blocks and blood specimens are collected for bio-banking and translational research.

After completion of study therapy, patients are followed up every 3 months.

ELIGIBILITY:
* Histologically proven grade II or grade III astrocytoma, oligodendroglioma or oligoastrocytoma according to the WHO 2007 at initial diagnosis.
* Demonstrated absence of 1p/19q co-deletion according to local diagnosis.
* Availability of biological material for central review processes and translational research projects
* First recurrence after initial treatment with either radiotherapy and/or chemotherapy.
* Enhancing recurrence on MRI scan.
* For non operated patients, recurrent disease must be at least one bi-dimensionally measurable contrast-enhancing lesion with clearly defined margins by MRI scan, with minimal diameters of 10 mm, visible on 2 or more axial slices 5 mm apart, based on MRI scan done within two weeks prior to start of randomisation.
* Stable or decreasing dosage of steroids for 7 days prior to the baseline MRI scan.
* No more than one line of chemotherapy (concurrent and adjuvant temozolomide chemotherapy is considered one line of chemotherapy)

  * If given, chemotherapy must have consisted of either temozolomide or PCV, and patients must be off chemotherapy treatment for more than 6 months without progression.
* No radiotherapy within the three months prior to the diagnosis of progression
* No radiotherapy with a dose over 65 Gy, stereotactic radiosurgery or brachytherapy unless the recurrence is histologically proven
* No current or recent (within 4 weeks before randomization) treatment with another investigational drug
* No prior treatment with Bevacizumab or other VEGF inhibitors or VEGF-Receptor signaling inhibitors
* No invasive procedures (surgical resection, open biopsy, significant traumatic injury or any other major surgery involving entry into a body cavity) within 4 weeks prior to randomization, or anticipation of the need for major surgery during the course of the study treatment.
* No core biopsy (excluding intracranial biopsy) or other minor surgical procedure within 7 days prior to randomization. Placement of a central vascular access device (CVAD) if performed at least 2 days prior to bevacizumab administration is allowed.
* Patient may have undergone surgery for recurrence. If operated, residual and measurable disease after surgery is not required but histology must have confirmed the recurrence. Craniotomy or intracranial biopsy site must be adequately healed free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of randomisation.
* No previous other malignancies, except for any previous malignancy which was treated with curative intent more than 5 years prior to randomisation, and except for adequately controlled limited basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix
* Absence of any cardiovascular disorder, including but not limited to:

  * No history of myocardial infarction, unstable angina within 6 months prior to randomisation
  * No "New York Heart Association" (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication.
  * No significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomisation
  * No prior history of hypertensive crisis or hypertensive encephalopathy
  * No inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 m Hg)
* Absence of any thrombotic or hemorrhagic event, including but not limited to:

  * No evidence of recent hemorrhage on MRI of the brain. However, patients with clinically asymptomatic presence of hemosiderin, resolving hemorrhagic changes related to surgery, and presence of punctate hemorrhage in the tumor are permitted entry into the study
  * No history or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
  * No arterial or venous thrombosis ≤ 12 months prior to randomization
  * No history of stroke or TIAs within 6 months prior to randomization
  * No history of pulmonary haemorrhage/haemoptysis ≥ grade 2 according to the NCI-CTCAE version 4.0 criteria within 1 month prior to randomization
  * Absence of current or recent (within 10 days of first dose of Bevacizumab) use of aspirin (> 325 mg/day) or other NSAID with anti-platelet activity or treatment with dipyramidole, ticlopidine, clopidogrel or cilostaz.
  * International normalized ratio (INR) > 1.5 ULN and activated partial thromboplastin time (aPTT) > 1.5 × the ULN. Patients using full-dose anticoagulants at baseline are excluded from the study; but prevention of thrombosis with low-dose anticoagulant is allowed
* Absence of known hypersensitivity

  * to any part of the Bevacizumab or Temozolomide formulations.
  * to Chinese hamster ovary cell products or other recombinant human or humanized antibody.
* No underlying or previous conditions that could interfere with treatment, including but not limited to:

  * No history of intracranial abscess within 6 months prior to randomisation
  * No clinically serious (as judged by the investigator) non-healing wounds, active skin ulcers or incompletely healed bone fracture.
  * No history of active gastroduodenal ulcer(s).
  * No history of abdominal fistula as well as non-GI fistula, gastrointestinal perforation or intraabdominal abscess within 6 months prior to inclusion.
  * No evidence of active infection requiring hospitalization or antibiotics, within 2 weeks prior to randomisation.
  * No other diseases, interfering with follow up.
* Normal hematological functions: neutrophils ≥ 1.5 x 109 cells/l, platelets ≥100 x 109 cells/l and Hb ≥ 6.2 mmol/l (9.9 g/dl).
* Normal liver function: bilirubin < 1.5 x upper limit of the normal range (ULN), alkaline phosphatase and transaminases (ASAT) < 2.5 x ULN, INR < 1.5 ULN.
* Normal renal function: calculated (Cockcroft-Gault) or measured creatinine clearance > 30 mL/min; Urine dipstick for proteinuria < 2+. Patients with ≥2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hours urine collection and must demonstrate ≤1 g of protein/24 hr.
* Age ≥ 18 years
* WHO Performance status 0 - 2
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. In general, the decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal.

  * Post menopause is defined as: amenorrhea ≥ 12 consecutive months without another cause or for women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
  * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.
  * Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.
* Female patients within one year of entering the menopause as well as males must agree to use an effective non-hormonal method of contraception during the treatment period and for at least 6 months after the last study treatment.
* Female should not be breast feeding
* Absence of any psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule; such conditions should be assessed with the patient before randomization in the trial.
* Before patient randomization and study related procedures (that would not have been performed as part as standard care), written informed consent must be given according to ICH/GCP, and national/local regulations. Informed consent should also be given for biological material to be stored and used for future research on brain tumors.
* All indicated timelines and absolute values requested by the eligibility criteria must be adhered to. However, a maximum of +/- 10% of the reference value for laboratory parameters and a maximum of +/- 2 days for timelines may be acceptable. Discussion with Headquarters and study coordinator is encouraged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2011-02; Primary Completion 2017-01-19 (Actual); Study Completion 2017-09-24 (Actual)

PRIMARY OUTCOMES:
Probability of survival at 1 year | From the date of randomization up to the date of death, assessed up to 12 months
  Patients alive at 12 months

SECONDARY OUTCOMES:
Objective response rate and duration of response | From the date of randomization until disease progression
  Objective response includes best overall responses complete response and partial response
Progression-free survival | From the date of randomization until the date of objective progression or the date of patient's death whichever occurs first
Overall survival and survival at 24 months | From the date of randomization up to the date of death
Safety | After the first ten patients in each arm have completed the first two cycles or have stopped treatment, an interim safety review of those patients will be conducted.
Clinical/neurological deterioration-free survival | From the date of randomization until the date of neurological deterioration
Steroid use | At baseline and every 3 months untill lost to follow-up
Quality of life of patients and caregivers/relatives | At baseline and every 3 months untill lost to follow-up
Cognitive deterioration | At baseline and every 3 months untill lost to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. van Den Bent, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center; Ahmed Idbaih, Study Chair — CHU Pitie-Salpetriere
Locations (39):
- Austria (2):
  - Landesnervenklinik Wagner Jauregg, Linz
  - Medical University Vienna - General Hospital AKH, Vienna
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- France (9):
  - CHRU de Lille, Lille
  - CHU de Lyon - CHU Lyon - Hopital neurologique Pierre Wertheimer, Lyon
  - Assistance Publique - Hôpitaux de Marseille - Hôpital de La Timone, Marseille
  - CHU de Nice - Hopital Pasteur, Nice
  - CHU Pitie-Salpetriere, Paris
  - Institut Gustave Roussy, Paris
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
- Germany (5):
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum - Essen, Essen
  - Klinikum Der J.W. Goethe Universitaet, Frankfurt am Main
  - Universitaetsklinikum Heidelberg - UniversitaetsKlinikum Heidelberg - Head Hospital, Heidelberg
  - Universitaetskliniken Regensburg, Regensburg
- Ospedale Bellaria, Bologna, Italy
- Netherlands (6):
  - University Medical Center Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - Medisch Centrum Haaglanden - Westeinde, The Hague
  - Universitair Medisch Centrum - Academisch Ziekenhuis, Utrecht
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - UniversitaetsSpital Zurich - Division of Oncology, Zurich
- United Kingdom (12):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - University Of Dundee - Ninewells Hospital, Dundee
  - NHS Lothian - Western General Hospital, Edinburgh
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust - St. James's University Hospital, Leeds
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London
  - University College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Northern Centre For Cancer Care, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield
  - Royal Marsden Hospital - Sutton, Surrey, Sutton

REFERENCES:
- [Derived] Draaisma K, Tesileanu CMS, de Heer I, Klein M, Smits M, Reijneveld JC, Clement PM, de Vos FYF, Wick A, Mulholland PJ, Taphoorn MJB, Weller M, Chinot OL, Kros JM, Verschuere T, Coens C, Golfinopoulos V, Gorlia T, Idbaih A, Robe PA, van den Bent MJ, French PJ. Prognostic Significance of DNA Methylation Profiles at MRI Enhancing Tumor Recurrence: a Report from the EORTC 26091 TAVAREC Trial. Clin Cancer Res. 2022 Jun 1;28(11):2440-2448. doi: 10.1158/1078-0432.CCR-21-3725. PMID 35294545
- [Derived] van den Bent MJ, Klein M, Smits M, Reijneveld JC, French PJ, Clement P, de Vos FYF, Wick A, Mulholland PJ, Taphoorn MJB, Lewis J, Weller M, Chinot OL, Kros JM, de Heer I, Verschuere T, Coens C, Golfinopoulos V, Gorlia T, Idbaih A. Bevacizumab and temozolomide in patients with first recurrence of WHO grade II and III glioma, without 1p/19q co-deletion (TAVAREC): a randomised controlled phase 2 EORTC trial. Lancet Oncol. 2018 Sep;19(9):1170-1179. doi: 10.1016/S1470-2045(18)30362-0. Epub 2018 Aug 13. PMID 30115593
- [Derived] Ediebah DE, Reijneveld JC, Taphoorn MJ, Coens C, Zikos E, Aaronson NK, Heimans JJ, Bottomley A, Klein M; EORTC Quality of Life Department and Patient Reported Outcome and Behavioral Evidence (PROBE). Impact of neurocognitive deficits on patient-proxy agreement regarding health-related quality of life in low-grade glioma patients. Qual Life Res. 2017 Apr;26(4):869-880. doi: 10.1007/s11136-016-1426-z. Epub 2016 Oct 15. PMID 27744512